CLINICAL TRIAL: NCT03348098
Title: Tianjin Medical University Cancer Institute and Hospital
Brief Title: Clinical Study of Neoadjuvant Therapy With Apatinib and Paclitaxel in Local Advanced Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD TB001
Record Dates: First submitted 2017-11-09; First posted 2017-11-20 (Actual); Last update posted 2017-11-28 (Actual); Status verified 2017-09

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — apatinib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Apatinib Combined With Paclitaxel in Neoadjuvant Therapy of Locally Advanced Exploratory Research on Single-arm of TNBC
  Interventions: Drug: Apatinib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Apatinib — 500 mg, po, qd. 12weeks
  Other Names: YN968D1
Drug: Paclitaxel — drug: Paclitaxel ,80mg/m2, d1, Once a week , A total of 12 weeks; 3 weeks as a cycle
  Other Names: Taxol

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of apatinib in patient with TNBC

DETAILED DESCRIPTION:
NACT (Neoadjuvant chemotherapy) Increasingly widespread in clinical practice, there is still a substantial proportion of the patients NACT After failing to obtain ORR DCR , NACT Did not receive ORR DCR Patient access ORR DCR Patients have a higher risk of recurrence, and complete NACT The patient, the current standard therapy in the secondary stage of chemotherapy is no longer used, but non-ORR non-DCR After neo-adjuvant chemotherapy in patients with postoperative chemotherapy is worth exploring. Targeted drugs refer to interfere with tumor specific molecular processes and achieve inhibit or block the progression of drugs, its functioning is based on normal cells and tumor cells, differences, which makes the target specificity and side effects of the drug. Target drug is a pioneer in precision treatment of its interpretation of the individualized treatment based on the standard treatment. NCCN guidelines recommend paclitaxel in neoadjuvant chemotherapy is NACT first-line choice. At the Apatinib for dasatinib therapy in previous studies of breast cancer has a high level of performance, the Apatinib for dasatinib combined with paclitaxel in neoadjuvant therapy for breast cancer efficacy and safety is better than traditional treatments, is worthy of question.

ELIGIBILITY:
Inclusion Criteria:

1. patients between18 and 75 Years old;
2. patients with locally advanced breast cancer (TNM periodization:T is equal to or greater than 2,N is equal to 1,M is equal to 0)
3. clear for immunohistochemical is that: estrogen receptor-negative (ER-), progesterone receptor-negative (PR-), the human epidermal growth factor receptor 2 is Negative ( IHC Her-2 0/+ , If ER- 、 PR- But Her-2 ++ , You need to do FISH/CISH Testing confirmed that Her-2 Amplification is negative);
4. The ECOG score is between 0 to 2 points;
5. The expected lifetime is ≥3 months;
6. Major organ function is normal, that meet the following criteria:

   1. Blood test standards subject to:

      HB≥90 g/L ;

      ANC≥1.5×109 /L ;

      PLT≥100×109 /L ;
   2. Biochemical examination must meet the following criteria:

   TBIL≤1.5xULN ( upper limit of normal value ) ;

   ALT AST≤2.5×ULN ;

   Serum Cr≤1.5×ULN And endogenous creatinine clearance rate ≥50 mL/min (Cockcroft-Gault formula ) ;
7. the women of childbearing age must do the pregnancy test ( serum or urine ) within 7 days when they are included in the trial, And the result was negative, and during the trial and at the time of giving experimental drugs after 8 weeks using the appropriate methods of contraception;
8. no difficulty in swallowing, swallowing oral medications;
9. the participants volunteered to join this study should sign the informed consent forms, have better compliance, work in with the follow-up

Exclusion Criteria:

1. patients with pregnancy or lactation;
2. inflammatory breast cancer patients;
3. patients with several factors affecting medication (for example, inability to swallow, such as nausea, vomiting, chronic diarrhea, and bowel obstruction);
4. injury or pathologic fracture;
5. people with high blood pressure and antihypertensive drug treatment could not be reduced to within the normal range (systolic >140 mmHg, diastolic pressure >90 mmHg) ;
6. with ⅱ grade myocardial ischemia, poor control of arrhythmias or myocardial infarction (including QTc interval men ≥450 Ms, female ≥470 Ms);
7. according to NYHA standard ⅲ~ⅳ -class heart insufficiency or heart ultrasound: LVEF(left ventricular ejection fraction) <50%;
8. the past 6 months have gastrointestinal bleeding within history or definite gastrointestinal bleeding, such as: risk of bleeding oesophageal varicose ulcer lesions, fecal occult blood, local activities ≥ (++) Into groups; such as the fecal occult blood (+), requires endoscopy;
9. prior to participating in the study of 28 days abdominal fistula, perforation of the gastrointestinal tract and abdominal abscesses;
10. positive patients of urinary protein (urine protein 2+ or above, or 24 -hour urine protein > 1.0g);
11. distant metastasis of patients with symptoms or are not controlled;
12. expected lifetime < 3 months;
13. into the group before 28 days to accept other anticancer treatment;
14. other information: dysfunction of blood coagulation (INR>1.5 or prothrombin time ( PT )> ULN+4 Seconds); Anticoagulant therapy are receiving antithrombotic or infection who needed intravenous antibiotics; previously receiving bevacizumab treatment or other anti- VEGF TKI Drug treatment, with a second tumor (except basal cell carcinoma and cervical carcinoma in situ);
15. a history of immunodeficiency, including HIV testing positive, or suffer from other acquired, congenital immune deficiency disease or have a history of organ transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-09-06 (Actual); Primary Completion 2018-07-06 (Estimated); Study Completion 2018-12-06 (Estimated)

PRIMARY OUTCOMES:
ORR | ten months
  objective response rate

SECONDARY OUTCOMES:
DCR | ten months
  disease control rate
pCR | ten months
  pathologic complete response
DFS | ten months
  disease free survival
Incidence of Treatment-Emergent Adverse Events [Safety] | ten months
  incidence of participants with treatment-related adverse events as assessed by NCI CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: Hong MD Liu, Study Chair — study principal investigator
Locations (1):
- TianJin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: Undecided
the plan to share IPD is under consideration